CLINICAL TRIAL: NCT04721834
Title: Efficacy of Low-Intensity Extracorporeal Shockwave Therapy in Treatment of Erectile Dysfunction - A Randomized Controlled Trial With Sham Therapy
Brief Title: LI-ESWT Versus Sham Therapy in Men With ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, CHENG Kwun-Chung, Associate Consultant, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEC-ESWT-RCT
Record Dates: First submitted 2020-10-15; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: During treatment for the placebo arm, a sham probe will be used which will produce a noise mimicking active treatment.
  Subjects would be blinded from randomization, treatment, until the end of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity ESWT (Active Comparator): Patient would be positioned in a supine position. Shockwaves would be delivered to the stretched penis at proximal, mid and distal penile shaft and bilateral crura of penis. (Energy: 0.1-0.25 mJ/mm2; 3000pulses per session; Frequency 3Hz) Treatment consists of 6 sessions over 5 weeks in total. It would be a twice-weekly treatment with one-week interval of resting period. Patient would be discharged home after each treatment session.
  Interventions: Device: Low-intensity Extracorporeal Shockwave Therapy
- Sham ESWT (Sham Comparator): Sham therapy would be given with a modified probe which no shockwave would be emitted. A working noise would still be generated which mimicked active treatment.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Low-intensity Extracorporeal Shockwave Therapy — Low intensity shockwave energy would be delivered to stimulate angiogenesis in corporal tissue. Therapy would be delivered through a linear probe in 6 sessions. It would be conducted as a day procedure.
  Arms: Low-intensity ESWT
Device: Sham Therapy — Same device as the active treatment arm would be used, with the addition of sham probe which block all shockwaves.
  Arms: Sham ESWT

SUMMARY:
Hong Kong has an aging population. By the year of 2036, more than 30% of our population will be older than 65 years old1. Aging in male has been shown to correlate with the risk of erectile dysfunction(ED). The demand in ED treatment is expected to increase.

Several ED treatment options are available, ranging from oral or intracavernosal drug treatments, to vacuum erection therapy or even penile prosthesis implantation. However, none of these treatment are curative nor rectify the pathophysiology of ED. Low-intensity extra-corporeal shockwave therapy(LI-ESWT) has been introduced since 2010 for treatment of ED. The first randomized-controlled trial by Vardi et al. had proved the efficacy of ESWT in improving the International Index of Erectile Function(IIEF) score3. The International Index of Erectile Function-Erectile Function domain score(IIEF-EF) was significantly greater in the treatment group compared with the sham therapy group. The efficacy of LI-ESWT was also confirmed in meta-analyses. Nonetheless, the available studies were criticized for the variations in shockwave generators, energy parameters and treatment protocol. Most studies used focused electrohydraulic machines, did not include NPT as part of the outcomes assessment, and only reported the short-term outcomes.

Currently LI-ESWT machine was used in few Hong Kong public hospitals for the treatment of erectile dysfunction. In KEC, few pilot cases have been done using the linear LI-ESWT machine. No adverse events were seen. Local published data is lacking. Yee et al. has published a double-blinded randomized placebo-controlled trial on LI-ESWT in 20144. Using an electrohydraulic machine with a focused shockwave source, they concluded no significant differences in IIEF-EF and Erectile Hardness Score(EHS) between treatment and sham therapy after 13 weeks of treatment. In subgroup analysis significant improvement was noted in men with severe baseline erectile dysfunction (LI-ESWT IIEF-EF improvement: 10.1 ± 4.1 vs sham therapy IIEF-ED domain improvement: 3.2 ± 3.3; P = 0.003). There were several limitations in this study. These include the small number of participants included in the subgroup analysis (ranges from 18 to 21 men in each subgroups), the lack of physical measurement of erectile function. The percentage of patients with 5 points or more IIEF-EF improvement and the Erection Hardness Score(EHS) were also not reported. They have also used an old design with focused energy source, instead of the linear energy source.

In light of the limitations of the previous international and local studies, the investigators plan to investigate the efficacy of a linear electromagnetic LI-ESWT machine in men with moderate and severe ED. In addition, the intermediate-term outcomes would be studied, in terms of patients-reported erection scores and nocturnal tumescence and rigidity measurement.

DETAILED DESCRIPTION:
Objectives

1. To investigate the efficacy and safety of LI-ESWT in treatment of moderate and severe ED
2. To investigate the effect of LI-ESWT on nocturnal penile tumescence and rigidity.

Research Plan and Methodology

1. Study Design This is a prospective, two-centre randomized controlled trial involving United Christian Hospital and Tseung Kwan O Hospital. The study will be conducted in accordance with the Declaration of Helsinki and the International Conference on Harmonisation, Good Clinical Practice Guidelines (ICH-GCP). This RCT will be registered with ClinicalTrials.gov.
2. Patient selection and recruitment Patients would be recruited in the urology outpatient clinics. Subjects who fulfilled selection criteria would be counselled to participate in the study. Written consent would be obtained.
3. Randomisation, allocation concealment and blinding Patients are randomised to either LI-ESWT or sham therapy in a ratio of 1:1. Randomisation is performed with a random number table. The designated operator who perform the procedure is not blinded. Patients were blinded throughout the procedures, during clinical follow-up and data analysis.
4. Study Intervention Patients would undergo a 4-week washout period of oral phosphodiesterase inhibitors after recruitment. Severity of ED would be assessed by the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) & International Index of Erectile Function (IIEF-5) questionnaires and Erection Hardness Score(EHS) after the washout. Nocturnal penile tumescence (NPT) and rigidity would be measured by the Rigiscan at the night prior to the first treatment.

   All procedures would be performed by a designated nurse consultant(co-investigator) in an office setting using an electromagnetic linear shockwave machine. The nurse consultant has received overseas andrology training, as well as on-hand machine operation training by ESWT product specialist. Patient would be positioned in a supine position. Shockwaves would be delivered to the stretched penis at proximal, mid and distal penile shaft and bilateral crura of penis. (Energy: 0.1-0.25 mJ/mm2; 3000pulses per session; Frequency 3Hz) Treatment consists of 6 sessions over 5 weeks in total. It would be a twice-weekly treatment with one-week interval of resting period. Patient would be discharged home after each treatment session. Sham therapy would be given with a modified probe which no shockwave would be emitted. A working noise would still be generated which mimicked active treatment.
5. Post-procedure management Clinical assessment would be conducted at week 4, week 26 and week 52 after completion of treatment. NPT would be measured at week 4. At all follow-up the IIEF-EF and EHS would be assessed. Any complications would be assessed and documented according to Clavien-Dindo classification.
6. Sample Size Calculation In a recent meta-analysis, the mean improvement in IIEF-EF was 4.23. At 5% significance level and 80% power, 33 subjects were needed in each treatment and sham group (Total 66 subjects). Overall 84 subjects would be recruited with 20% of drop out expected (i.e. 42 subjects in each group).
7. Study Period The expected study period would last for 44 months, including 30 months of subject enrolment, 2 months of treatment and 12 months of follow-up.
8. Statistical Analysis The results would be analysed according to intention-to-treat principle. Mann-whitney U test would be used to study the IIEF-EF results, as well as all other non-parametric continuous variables in secondary outcomes. Chi-square test would be used for categorical variable, independent samples t-test would be used for parametric continuous variable.

Ethical Concern All identifiable personal data will be anonymised and will follow the HA policy on handling of patient data privacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years old
* ED > 6 months
* Stable heterosexual relationship > 6 months
* Sexual Health Inventory for Men (SHIM) score <= 16
* Suboptimal response after first line phosphodiesterase type 5 inhibitor treatment

Exclusion Criteria:

* Penile anatomical abnormality
* History of pelvic radiotherapy
* History of radical prostatectomy
* History of penile implantations
* Neurological diseases
* Hypogonadism or on anti-androgen therapy
* Unstable psychiatric conditions or under active psychiatric treatment

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male subjects are eligible.
Enrollment: 84 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in International Index of Erectile Function - Erectile Function Domain (IIEF-EF) score | One month after treatment, compared with pre-op level
  Validated questionnaire in assessing the erectile function over the past 4 weeks Minimum value - 1 Maximum values - 30 Higher scores represent a better outcome

SECONDARY OUTCOMES:
Erection Hardness Score (EHS) | At week 4, 26 and 52 after treatment
  Hardness score of penis. Minimum value is 1, maximum is 4. Higher score represents better erection hardness.
Percentage of patients with 5-points International Index of Erectile Function - Erectile Function Domain improvement | At week 4, 26 and 52 after treatment
  The percentage(%) of patients with 5 points or more International Index of Erectile Function - Erectile Function improvement compared with pre-study baseline level.
Percentage of patients with Erection Hardness Score improved to 3 or above | At week 4, 26 and 52 after treatment
  The percentage(%) of patients with Erection Hardness Score improved to 3 or above.
Frequency of nocturnal erections | At week 4 and 52 after treatment
  A non-invasive ambulatory diagnostic machine Rigiscan would be used to provide an objective measure of the frequency of nocturnal erections at night. (number of erections during sleeping)
Duration of nocturnal erections | At week 4 and 52 after treatment
  A non-invasive ambulatory diagnostic machine Rigiscan would be used to provide an objective measure of the duration of nocturnal erections.(Time in seconds)
Change in nocturnal penile tumescence | At week 4 and 52 after treatment
  A non-invasive ambulatory diagnostic machine Rigiscan would be used to provide an objective measure of the change in penile girth at penile base and penile tip during nocturnal erections.(in cm)
Complications after the procedure | Within 4 weeks after treatment
  Number of participants reported penile pain or urethral bleeding during treatment or within 4 weeks after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kwun Chung CHENG, FRCS, Principal Investigator — Hospital Authority, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Yee CH, Chan ES, Hou SS, Ng CF. Extracorporeal shockwave therapy in the treatment of erectile dysfunction: a prospective, randomized, double-blinded, placebo controlled study. Int J Urol. 2014 Oct;21(10):1041-5. doi: 10.1111/iju.12506. Epub 2014 Jun 17. PMID 24942563
- [Background] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Background] Campbell JD, Trock BJ, Oppenheim AR, Anusionwu I, Gor RA, Burnett AL. Meta-analysis of randomized controlled trials that assess the efficacy of low-intensity shockwave therapy for the treatment of erectile dysfunction. Ther Adv Urol. 2019 Mar 29;11:1756287219838364. doi: 10.1177/1756287219838364. eCollection 2019 Jan-Dec. PMID 30956690

DOCUMENTS (1):
  • Informed Consent Form (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT04721834/ICF_000.pdf